CLINICAL TRIAL: NCT04300049
Title: Effect of Physiologic Hyperglucogonemia on Adipocyte Metabolism
Acronym: Glucagon
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: South Texas Veterans Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HSC20170682H
Record Dates: First submitted 2020-03-05; First posted 2020-03-09 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Insulin Sensitivity
Keywords: glucagon; Lipolysis
MeSH Terms: conditions — Insulin Resistance | interventions — Glucagon; Sodium Chloride; Saline Solution

STUDY DESIGN:
Intervention Model Description: single arm before and after glucagon vs. saline
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Change in Glycerol Ra (Experimental): The difference in rate of lipolysis (glycerol Ra) during the basal state (-120 -0 minute) between subjects receiving glucagon and saline represents the change in whole body lipolysis caused by glucagon.
  Interventions: Drug: Glucagon Infusion; Other: Saline

INTERVENTIONS:
Drug: Glucagon Infusion — Study participants will receive glucagon infusion (6ug/kg/min for 12 hours) 12 hours.
  Other Names: IV Glucagon
Other: Saline — Study participants will receive saline infusion for 12 hours.
  Other Names: Normal saline

SUMMARY:
Purpose/Objectives: To investigate the effect of hyperglucagonemia on insulin action, particularly on adipose tissue.

Research Design/Plan: Normal glucose tolerant subjects will be studied. Study subjects will receive a continuous glucagon infusion for 12 hours. Following glucagon infusion, subjects will receive prime-continuous tracer infusions for additional 4 hours to measure adipocyte metabolism. Within 6-8 weeks, subjects will return for a repeat study with normal saline as a control group.

Methods: All subjects will have an oral glucose tolerance test prior to participation to confirm they are normal glucose tolerant. Subjects will be admitted to the CRC at 4 PM and will receive a continuous glucagon for 12 hours. At 6 AM on the following morning, subjects will receive prime-continuous tracer infusions of the following for 4 hours (14C-glycerol, 3-3H glucose, and D2O). At 10 AM continuous indirect calorimetry will be performed to determine rates of energy expenditure and glucose/lipid oxidation for 40 minutes. At 6 AM a surgical biopsy of abdominal adipose tissue will be performed for measurement of adipocyte metabolism. At 8 AM, the study team will infuse insulin/glucose to test for insulin sensitivity.

Clinical Relevance: The results of this study will help the study team to further understand the pathophysiology of metabolic disturbances that is induced by hyperglucagonemia in type 2 diabetes patients.

DETAILED DESCRIPTION:
Visit 1 Screening: All subjects will be performed indirect calorimetry to determine rates of energy expenditure and glucose/lipid oxidation for 40 minutes prior to all other procedures to obtain a fasting calorimetry. Subjects then will have a 75 gram oral glucose tolerance test to document the presence of normal glucose tolerance. Blood will be drawn at -30, -15, 0 and at 15, 30, 45, 60, 90 and 120 minutes thereafter for the determination of plasma glucose, insulin, C-peptide, glucagon, FFA, glycerol, GLP-1 and GIP concentrations. The total amount of blood to be taken during the OGTT is 148 ml or about 10 tablespoons. Participants will also undergo a total body fat (DXA) and hepatic fat content (MRS). Subjects will also have a routine physical exam, an ECG, weight, height, vitals and collection of prior medical history. The study team will also check blood glucose (sugar) and blood lipid (fat) levels. The total amount of blood that we will take for the screening blood tests, HbA1c, lipid, and other blood tests is 34 ml or about 2 1/3 tablespoons.

Visit 2 Adipose Tissue Metabolism Measurement: Subjects (n=12) will be admitted to the CRC at 4 PM on the day prior to study and received a standardized, weight maintaining diet containing 50% CHO: 30% fat: 20% protein. At 6 PM subjects will receive a continuous glucagon (3 ng/kg.min, N=6) or glucagon (6 ng/kg.min, N=6) for 12 hours. Subjects will remain fasting after 10 PM. Samples for glucagon, FFA, insulin and C-peptide will be collected at 1700, 1730, 1800, 1900, 2100, 2300, 0100, 0300, and 0500 hours.

At 6 AM on the following morning subjects will receive prime-continuous tracer infusions of the following for 4 hours (see figure 1):

(i) 14-C-glycerol (prime = 30 µCi; continuous infusion = 0.3 µCi/min) for determination of total body rate of lipolysis.

(ii) 3-3H-glucose (prime = 40 µCi; continuous infusion = 0.4 µCi/min) for determination of rates of total body glucose appearance and disappearance.

(iii) D2O (5 g/kg fat free mass at 9 PM orally) to determine the rate of de novo lipogenesis.

At 6 AM a surgical biopsy of subcutaneous abdominal adipose tissue will be performed for measurement of hormone sensitive (HSL) lipase activity, AMPK activity, and serine phosphorylation of HSL (see Figure 2), FGF-21, FAP, Beta-klotho. Insulin signaling (IR/IRS-1 tyrosine phosphorylation, PI-3 kinase activity, Akt) molecules, GLUT4, markers of inflammation (IkB, NF-kB, T4R4TLR4, JNK, p38 MAPK, M2/M1 macrophages, IL-1, IL-6, TNF alpha, MCP-1) also will be measured on the fat biopsy. Lipidomic analysis to quantitate the amount of and type of fat in the adipose tissue biopsy also will be performed. After surgical biopsy of adipose tissue, starting the tracer equilibration (6AM) blood will be drawn every 15-30 minutes for 4 hours (6-10 AM) for substrate (glucose, FFA, glycerol, triglycerides), hormone (glucagon, insulin, C-peptide, GLP-1, GIP, adiponectin, leptin, FGF21 [active and total], FAP [degrading enzyme]), radioisotope (14-C-glycerol and 3-3H glucose) specific activity. Participants will place their hand in a transparent plastic thermo-regulated box heated to 50-60°C (122-140°F) to ensure good blood flow to the hand. Pasma samples for radioisotope activity (background) will be obtained at 6 AM. At 9 AM continuous indirect calorimetry will be performed to determine rates of energy expenditure and glucose/lipid oxidation for 40 minutes.

The glucagon infusion will be continued through the 4-hour tracer infusion (i.e. 6AM-10AM). At the end of the glucagon infusion (~10 AM) a repeat measurement of hepatic fat content will be obtained. A total of 366 ml of blood will be drawn.

At 8 AM the insulin sensitivity test will be done during the last two hours of the tracer infusion. During the 2 hours of the insulin sensitivity test, the insulin (60 mU/m2 ⋅ min) and glucose will be given through the catheter in the vein in the subject's arm to determine rates of whole-body insulin sensitivity. There are no expect adverse reactions to be experienced by the subjects during both infusions.

ELIGIBILITY:
Inclusion Criteria:

1. Fasting Glucose < 100 mg/dl
2. HbA1C < 5.7%
3. 2-h OGTT value < 140 mg/dl
4. Good general Health as determined by medical history, physical exam, screening lab tests, urinalysis, and EKG.
5. Weight Stable (±3 lbs) over the preceding 3 months
6. ages from 18-50
7. Male/Female
8. BMI from 23-28 kg/m2 -

Exclusion Criteria:

1. Subjects who participate in an excessively heavy exercise program.
2. Subjects taking any medication known to affect glucose tolerance will be excluded.
3. Cannot be pregnant
4. Hyper sensitive to glucagon

   -

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
the rate of glycerol turnover | 12 hours after the infusion
  effect of glucagon infusion on whole body lipolysis,

CONTACTS AND LOCATIONS:
Overall Officials: Ralph DeFronzo, MD, Principal Investigator — University of Texas Health San Antonio
Locations (2):
- United States (2):
  - South Texas Veterans Health Care Center, San Antonio, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No